CLINICAL TRIAL: NCT04617158
Title: Comparison Between Immediate Versus Late Postoperative Adjustable Eye Muscle Surgery
Brief Title: Comparing Adjustable Sutures Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sahar T A Abdelaziz, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Minia University 2020
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Strabismus, Comitant
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early adjustable suture surgery (Active Comparator): Suture adjustment after 2 hours of surgery
  Interventions: Procedure: Adjustable strabismus surgery
- Late adjustable suture surgery (Active Comparator): Suture adjustment after 24 hours of surgery
  Interventions: Procedure: Adjustable strabismus surgery

INTERVENTIONS:
Procedure: Adjustable strabismus surgery — Adjustable surgery will be done using sliding nose technique using fornix approach

SUMMARY:
Adjustable suture surgery will be done in patients with horizontal strabismus comparing the time of adjustment

DETAILED DESCRIPTION:
Forty patients will be equally divided into two groups and time of adjustment of the suture will be compared as regards efficacy and pain tolerance

ELIGIBILITY:
Inclusion Criteria:

* More than 16 years old patients Comitant esodeviation and exodeviation 15-45 prism diopters Cooperative patients

Exclusion Criteria:

* Patients with previous strabismus surgery Patients with oblique deviations

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Alignment of the strabismus | 3 months
  Percentage of patients with successful postoperative alignment using prism cover test for measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sahar TA Abdelaziz, MD, Principal Investigator — Faculty of Medicine, Minia University
Locations (1):
- Faculty of Medicine- Minia University, Minya, Egypt